CLINICAL TRIAL: NCT06890832
Title: A Phase-2, Open-label, Randomized, Parallel-Group, Three-Arm Study to Assess Efficacy and Safety of Cabazitaxel Lipid Tablet in Combination with Prednisone for the Treatment of Adult Men with Metastatic Castration-Resistant Prostate Cancer Previously Treated with a Docetaxel-containing Treatment Regimen
Brief Title: A Study to Investigate Efficacy and Safety of Different Dose Regimen of Oral Cabazitaxel Tablet in Adult Participants with Prostate Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jina Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0128-23
Record Dates: First submitted 2025-03-17; First posted 2025-03-24 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Metastatic Castration-resistant Prostate Cancer, MCRPC
MeSH Terms: interventions — cabazitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm 1 (Experimental)
  Interventions: Drug: 50 mg cabazitaxel
- Arm 2 (Experimental)
  Interventions: Drug: 100 mg cabazitaxel
- Arm 3 (Experimental)
  Interventions: Drug: 200 mg cabazitaxel

INTERVENTIONS:
Drug: 50 mg cabazitaxel — 50 mg cabazitaxel to be taken every week for 6 cycles (3 doses per cycle), 10 mg prednisone to be taken daily till end of cycle 6
  Arms: Arm 1
Drug: 100 mg cabazitaxel — 100 mg cabazitaxel to be taken every week for 6 cycles (3 doses per cycle), 10 mg prednisone to be taken daily till end of cycle 6
  Arms: Arm 2
Drug: 200 mg cabazitaxel — 200 mg cabazitaxel to be taken every 3-week for 6 cycles (1 dose per cycle), 10 mg prednisone to be taken daily till end of cycle 6
  Arms: Arm 3

SUMMARY:
A total of 75 participants will be enrolled in the study, with 25 participants allocated per intervention group. In Group 1, participant will take 50 mg cabazitaxel every week for 6 cycles (3 doses per cycle), 10 mg prednisone daily till the end of cycle 6. In Group 2, participant will take 100 mg cabazitaxel every week for 6 cycles (3 doses per cycle), 10 mg prednisone daily till the end of cycle 6. In Group 3, participant will take 200 mg cabazitaxel every 3 weeks for 6 cycles (1 doses per cycle), 10 mg prednisone daily till the end of cycle 6.

The study comprises three phases: a 21-day screening phase, an 18-week intervention phase starting on Day 1 (baseline), and a post-intervention follow-up phase lasting up to 12 months from Day 1. The total duration of participation for each individual will be approximately one year.

Key efficacy assessments include CT scans/MRI, bone scans, PSA, ALP, LDH, symptomatic skeletal events, and pain evaluations. Key safety assessments encompass the monitoring of adverse events (AEs), ECOG performance status, physical examinations, vital sign measurements, clinical laboratory tests, peripheral neuropathy evaluation, 12-lead ECG, and echocardiogram (ECHO) assessments.

Pharmacokinetic parameters will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Must sign an ICF indicating that the participant understands the purpose of, and procedures required for the study.
2. Male participant ≥18 years of age at the time of signing the informed consent.
3. Participant must have histological pathological, and/or cytological confirmation of adenocarcinoma of the prostate.
4. Evidence of metastatic disease.
5. Participant must be previously treated with a docetaxel-containing regimen (at least 3 cycles) for the treatment of prostate cancer (including locally confined inoperable disease that cannot be treated with definitive intent) and/or CRPC. Docetaxel administration in combination with androgen deprivation therapy (ADT) with or without next-generation AR-targeted therapy (abiraterone acetate, enzalutamide, or and next generation targeted agents Darolutamide, apalutamide) in metastatic hormone-sensitive disease is considered a prior docetaxel exposure.
6. Progressive disease prior to screening by PSA or imaging per PCWG3 criteria during or following the direct prior line of therapy in the setting of medical or surgical castration.
7. Participant must be taking ADT with a gonadotropin-releasing hormone (GnRH) analogue or bilateral orchiectomy (i.e., surgical or medical castration) confirmed by testosterone level ≤1.73 nmol/L (50 ng/dL) at the screening visit.
8. Participant must be eligible for treatment with cabazitaxel per the locally approved prescribing information.
9. ECOG PS grade of 0-2. ECOG PS 2 must be related to prostate cancer, not to other comorbidities.
10. Estimated life expectancy of ≥6 months as assessed by the investigator.
11. Participant has recovered from AEs (baseline or ≤ CTCAE Grade 1) due to prior anticancer therapy, unless AE(s) is either clinically nonsignificant or stable on supportive therapy or do not constitute a safety risk to the participant as determined by the investigator.
12. Male participants are eligible to participate if they agree to the following during the intervention period and for at least 6 months after the last dose of study intervention:

    * Must agree not to plan to father a child or donate sperm for the purpose of reproduction. PLUS, either of the following:
    * Be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long-term and persistent basis) and agree to remain abstinent OR
    * Must agree to use contraception /barrier
13. Participant with adequate hematologic, liver and renal function.
14. Willing and able to adhere to the lifestyle restrictions specified in this protocol.

Exclusion Criteria:

1. Known allergies, hypersensitivity, or intolerance to any of the study interventions, or components/ excipients thereof (refer to the IB), or drug or other allergy that, in the opinion of the investigator, contraindicates participation in the study.
2. Contraindications to the use of prednisone or medical ADT per locally approved prescribing information.
3. Previous treatment with cabazitaxel in any setting.
4. Had major surgical procedure or significant traumatic injury requiring general anaesthesia within 4 weeks or will not have fully recovered from surgical procedure prior to first dose of the study intervention; or has surgical procedure planned during the time the participant is expected to participate in the study.
5. Prior isotope therapy, whole pelvic radiotherapy or radiotherapy to >30% of bone marrow within 3 months prior to Baseline.
6. Symptomatic peripheral neuropathy Grade ≥2 (National Cancer Institute Common Terminology Criteria [NCI CTCAE] v.5.0).
7. Presence of hepatitis B surface antigen (HbsAg) at screening or within 3 months prior to first dose of investigational intervention.
8. Positive hepatitis C antibody test result at screening or within 3 months prior to starting investigational intervention.
9. Has known human immunodeficiency virus (HIV) seropositive status, or positive HIV antibody test at screening.
10. History of malignancy (except for prostate cancer) within the past 5 years except if the participant has undergone potentially curative therapy with no evidence of that disease recurrence for at least 3 years since initiation of that therapy.
11. • Current or chronic history of liver disease. This includes [but is not limited to hepatitis virus infections, drug- or alcohol-related liver disease, non-alcoholic steatohepatitis, autoimmune hepatitis, hemochromatosis, Wilson's disease, α-1 antitrypsin deficiency, primary biliary cholangitis, primary sclerosing cholangitis, or any other liver disease considered clinically significant by the investigator.

    • Known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
12. Participant with clinically significant current or recent (within the past 3 months before randomization [unless otherwise specified below]) cardiac conditions.
13. Known active CNS disease, except for treated stable asymptomatic CNS metastases.
14. Known Leptomeningeal disease.
15. Unmanageable concurrent bladder outflow obstruction or urinary incontinence.
16. Has an active infection requiring systemic therapy.
17. Spinal cord compression not definitively treated with surgical procedure and/or radiation, or previously diagnosed and treated spinal cord compression without evidence that disease has been clinically stable for ≥4 weeks prior to Baseline.
18. Received an investigational intervention or used an invasive investigational medical device within 30 days or 5 half-lives prior to the first dose of study intervention, whichever is longer.
19. Unable to swallow solid, oral dosage forms whole with the aid of water (participants cannot chew, divide, dissolve, or crush the investigational intervention) or and subjects with gastrointestinal disorders likely to interfere with absorption of the study medication.
20. Documented medical history of uncontrolled, clinically significant intercurrent medical condition(s) for which, in the opinion of the investigator, participation would not be in the best interest of the participant (e.g., compromise the well-being) or that could prevent, limit, or confound the protocol-specified assessments.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Radiographic progression-free survival (rPFS) | 12 months